CLINICAL TRIAL: NCT02387125
Title: A Phase 1b Study Evaluating the Safety, Tolerability and Immunogenicity of CMB305 (Sequentially Administered LV305 and G305) in Patients With Locally Advanced, Relapsed, or Metastatic Cancer Expressing NY-ESO-1
Brief Title: Phase 1b Safety Study of CMB305 in Patients With Locally Advanced, Relapsed, or Metastatic Cancer Expressing NY-ESO-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study did not meet the efficacy objective
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: V943A-001; IMDZ-C131 (Other: ImmuneDesign Protocol Number)
Record Dates: First submitted 2015-03-01; First posted 2015-03-12 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma; Melanoma; Non-small Cell Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Sarcoma; Melanoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — TLR4 agonist G100; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 Dose Escalation of CMB305 (Experimental): Patients with melanoma, NSCLC, ovarian cancer, or sarcoma will be enrolled. Patients will receive CMB305, a sequential regimen of LV305 and G305. Two cohorts are planned based on LV305 dose.
  Interventions: Biological: CMB305
- Part 2 Expansion of CMB305 (Experimental): Arm A will enroll up to 9 patients each with NSCLC or ovarian cancer, or up to 18 patients with the sarcoma subtypes, synovial sarcoma or MRCL. Arm B will enroll up to 9 additional patients with selected sarcoma subtypes to explore subcutaneous (SC) dosing of LV305 and G305 on the same schedule. Arm C will enroll up to 9 patients with synovial sarcoma or MRCL for treatment with CMB305 and with oral metronomic CPA. Arm D will enroll up to 9 patients with synovial sarcoma or MRCL at selected sites for treatment with CMB305 and IT G100. Arm E will enroll up to 6 patients with soft tissue sarcoma any subtype for treatment with a higher dose of CMB305 than previous arms.
  Interventions: Biological: CMB305; Biological: G100; Drug: Metronomic CPA

INTERVENTIONS:
Biological: CMB305
Biological: G100
  Arms: Part 2 Expansion of CMB305
Drug: Metronomic CPA
  Other Names: Cytoxan Tablets
  Arms: Part 2 Expansion of CMB305

SUMMARY:
This is a Phase 1b, open label, multi-center study of CMB305 (sequentially administered LV305 [a dendritic cell-targeting viral vector expressing the NY-ESO-1 gene] and G305 [NY-ESO-1 recombinant protein plus GLA-SE]) in patients with melanoma, sarcoma, ovarian cancer, or non-small cell lung cancer that express NY-ESO-1.

DETAILED DESCRIPTION:
This study is designed to investigate and examine the safety and immunogenicity of the combinatorial regimen called CMB305, where intradermal LV305 is administered sequentially with intramuscular G305 over three months. During Part 1, a dose escalation design will be utilized in patients with melanoma, NSCLC, ovarian cancer, or sarcoma. After completion of Part 1, the study will be expanded in Part 2 and will enroll patients with NSCLC, ovarian cancer, synovial sarcoma or myxoid/round cell liposarcoma. While this is an exploratory study to evaluate the safety, tolerability and immunogenicity of the CMB305 regimen, the study will also evaluate the safety and response to with oral metronomic CPA or intratumoral G100 in the context of CMB305.

CMB305 is a prime-boost vaccine approach against NY-ESO-1-expressing tumors, designed to generate an integrated, anti-NY-ESO-1 immune response in vivo via a targeted, specific interaction with dendritic cells.

G100 contains a potent synthetic small molecule toll-like receptor-4 (TLR-4) agonist, Glucopyranosyl Lipid A (GLA) that leverages the activation of both innate and adaptive immunity, including dendritic cells, in the tumor microenvironment to create an immune response against the tumor's preexisting diverse set of antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced, relapsed, and/or metastatic cancer
2. Tumor histology consistent with one of the following: In Part 1, Dose Escalation - melanoma, NSCLC, ovarian cancer (including fallopian tube carcinoma), or sarcoma (any subtype). In Part 2, Patient Expansion - NSCLC, ovarian cancer (including fallopian tube carcinoma), or the sarcoma subtypes, synovial sarcoma or myxoid/round cell liposarcoma
3. Tumor specimen positive for NY-ESO-1 expression by IHC and/or RT-PCR. At least one tumor must be accessible and patients must consent for biopsies in Arms C and D.
4. Inadequate response, relapse, and/or unacceptable toxicity with one or more prior systemic, surgical, or radiation cancer therapies, and for whom curative standard therapy is not an option (except patients with NSCLC who must have experienced either an inadequate response, relapse, and/or unacceptable toxicity with two or more prior systemic, surgical, or radiation cancer therapies)

6. ≥ 18 years of age 7. Life expectancy of ≥ 6 months per the investigator 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 9. ECG without evidence of clinically significant arrhythmia or ischemia 10. If female of childbearing potential (FCBP), willing to undergo pregnancy testing and agrees to use at least one highly effective or two effective contraceptive methods during the dosing period and for three months after last CMB305 injection 11. If male and sexually active with a FCBP, must agree to use highly effective contraception such as latex condom during the dosing period and for three months after last CMB305 injection

Exclusion Criteria:

1. Investigational therapy within 3 weeks prior to CMB305 dosing
2. Prior administration of other NY-ESO-1-targeting immunotherapeutics
3. Significant immunosuppression from:

   1. Concurrent, recent (≤ 4 weeks ago) or anticipated treatment with systemic corticosteroids at any dose, or
   2. Other immunosuppressive medications such as methotrexate, cyclosporine, azathioprine (antihistamines, non-steroidal anti-inflammatory drugs and aspirin permitted) or conditions such as common variable hypogamma-globulinemia or exposures such as large field radiotherapy
4. Cancer therapies, including chemotherapy, radiation, biologics or kinase inhibitors, G-CSF or GM-CSF within 3 weeks prior to the first scheduled CMB305 dosing
5. Psychiatric, other medical illness or other condition that in the opinion of the PI prevents compliance with study procedures or ability to provide valid informed consent
6. Significant autoimmune disease with the exception of alopecia, vitiligo, hypothyroidism or other conditions that have never been clinically active or were transient and have completely resolved and require no ongoing therapy
7. Myocardial infarction within 6 months of study initiation, active cardiac ischemia or New York Heart Association (NYHA) Grade III or IV heart failure
8. Inadequate organ function including:

   1. Marrow: Peripheral blood leukocyte count (WBC) < 3000/mm3, absolute neutrophil count ≤ 1500/mm3, platelets < 75000/mm3, or hemoglobin < 10 gm/dL
   2. Hepatic: alanine aminotransferase (ALT), and aspartate aminotransferase (AST) > 2.5 x ULN, total serum bilirubin > 1.5 x ULN (patients with Gilbert's Disease may be included if their total bilirubin is ≤3.0 mg/dL)
   3. Renal: Creatinine > 1.5x ULN
   4. Other: INR (prothrombin time ratio) or partial thromboplastin time (PTT) >1.5 x ULN
9. History of other cancer within 3 years (except non-melanoma cutaneous malignancies and cervical carcinoma in situ).
10. Active tuberculosis or recent (< 2 week ago) clinically significant infection or evidence of active hepatitis B, hepatitis C or HIV infection
11. For melanoma: Uveal melanoma or LDH >1.1 x ULN
12. Brain metastases considered unstable as:

    1. Without confirmed stability over 60 days in patients previously treated with prior surgery or radiation; OR
    2. Associated with symptoms and/or findings; OR
    3. Requiring corticosteroids or anticonvulsants in the prior 60 days
13. Pregnant, planning to become pregnant, or nursing
14. Known allergy(ies) to any component of CMB305 or CPA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
The nature, frequency and severity of adverse events (AEs) and laboratory abnormalities in subjects receiving CMB305 alone or in combination with oral metronomic CPA or G100 | Up to 5 years since first study injection
  To evaluate the safety and tolerability of CMB305 (sequential administered doses of LV305 and G305) alone or in combination with oral metronomic CPA or G100 in subjects with locally advanced, relapsed, or metastatic cancer expressing NY ESO 1

SECONDARY OUTCOMES:
Time to Progression | Up to 5 years since first study injection
  To evaluate clinical responses (by Immune-related Response Criteria (irRC) modified to use RECIST (v 1.1) measurement criteria), time to progression (TTP) and progression-free survival (PFS) as a preliminary assessment of clinical activity
Progression Free Survival | Up to 5 years since first study injection
  To evaluate clinical responses (by Immune-related Response Criteria (irRC) modified to use RECIST (v 1.1) measurement criteria), time to progression (TTP) and progression-free survival (PFS) as a preliminary assessment of clinical activity
Overall Survival | Up to 5 years since first study injection
  Overall survival (OS), time to progression (TTP), and progression-free survival (PFS) and descriptive tumor responses. Evaluation of response will be by RECIST (v1.1) modified to use irRC measurement criteria and by changes in markers of tumor burden
Humoral and cellular immune responses at selected sites, as measured by changes from baseline anti-NY-ESO-1 immunity | Approximately 14 weeks
  To evaluate the cellular and humoral immunogenicity of CMB305 alone or in combination with mCPA or G100 in patients

OTHER OUTCOMES:
To evaluate pre- and post-regimen blood samples for potential biomarkers of immunogenicity and clinical tumor response | Approximately 14 weeks
To evaluate available pre- and post-regimen tumor tissue for histologic, immunohistologic, and genomic markers following administration of CMB305 alone or in combination with mCPA or G100 | Approximately 14 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Sarcoma Oncology Center, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided